CLINICAL TRIAL: NCT01150877
Title: Study of High-dose Vitamin D Supplementation in Stage-4 Colorectal Cancer Patients
Brief Title: High Dose Vitamin D Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Lotte & John Hecht Memorial Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H10-00028
Record Dates: First submitted 2010-06-22; First posted 2010-06-25 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Colorectal Cancer
Keywords: Vitamin D; Vitamin D3; colon cancer; rectal cancer; Cholecalciferol
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Dietary Supplement (e.g., vitamins, minerals) (Experimental): Experimental arm is supplemented with high-dose of vitamin D.
  Interventions: Drug: Vitamin D
- No Intervention (No Intervention)

INTERVENTIONS:
Drug: Vitamin D — We propose to study high-dose, oral vitamin D supplementation, raising serum 25-hydroxy-vitamin D (25(OH)D) concentrations to 200 -250 nmol/L, in metastatic colorectal cancer patients with safety, tolerability and survival as the main outcome measurements. The dose is not pre-set and will depend on the individual subjects' serum 25(OH)D concentration. Subjects will be supplemented for 16 months with a daily oral dose, followed by a 12 months follow-up period.
  Arms: Experimental Dietary Supplement (e.g., vitamins, minerals)

SUMMARY:
The purpose of this study is to investigate the therapeutic effect and the safety of high-dose vitamin D supplementation in metastatic colorectal cancer patients. We propose to supplement metastatic (stage 4) colorectal cancer patients with oral doses of vitamin D to raise serum 25-hydroxy-vitamin D [25(OH)D] levels to the high normal range of 200-250 nmol/L. The primary objective of this study is to evaluate the metabolic consequences, including tolerability and toxicity, of prolonged, high-dose physiological vitamin D in patients with colorectal cancer. The secondary objective is to evaluate patient survival with regards to high-dose vitamin D supplementation.

Hypothesis:

Whereas low doses of vitamin D reportedly play a significant role in prevention of colorectal cancers, do much larger (pharmacological) doses of vitamin D have a significant therapeutic effect against the same kind of cancer?

DETAILED DESCRIPTION:
Metastatic (stage 4) colorectal cancer patients who were randomly assigned to the treatment arm of this study will be orally supplemented with high doses of vitamin D to achieve serum 25(OH)D concentrations of 200-250 nmol/L (80-100 ng/ml). Therefore, the supplementation dosage is not pre-set but will be determined on an individual basis. Vitamin D supplementation will be continued for 16 months, followed by a 12 month follow up period. Monthly monitoring of serum 25(OH)D and calcium levels will assure the safety of our treatment protocol. Subjects in the control arm of the study will be receiving standard cancer care at InspireHealth that includes supplementation with at least 2,000 International Units of vitamin D.

ELIGIBILITY:
Inclusion Criteria (We will recruit stage 4 (metastatic) colorectal cancer patients who are clients at InspireHealth):

* Age > 18
* Histologically confirmed colon or rectal cancer
* Known metastatic disease (stage-4) confirmed histologically or radiologically
* Life expectancy of >8 months
* May receive anti-neoplastic therapy at the discretion of their physician
* Stable metastatic disease defined as no change in systemic for the month before and the month after commencing study
* Signed informed consent

Exclusion Criteria(Stage 4 colorectal cancer patients):

* Pregnant / lactating women
* Known hypersensitivity to vitamin D
* Pre-existing renal stone disease based on history
* Pre-existing hypercalcemia
* Severe renal or hepatic dysfunction (≥ 2x of the upper normal range)
* granulomatous disease (TB and sarcoid)
* unable to give informed consent in English (translations of study documents in languages other than English will not be provided)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-04-23 (Actual); Study Completion 2014-04-23 (Actual)

PRIMARY OUTCOMES:
The metabolic consequences, including tolerability and toxicity, of prolonged, high-dose physiological vitamin D in patients with colorectal cancer. | After 16 months of intervention
The metabolic consequences, including tolerability and toxicity, of prolonged, high-dose physiological vitamin D in patients with colorectal cancer. | After 12 months of follow-up

SECONDARY OUTCOMES:
Patient survival with regards to high-dose vitamin D supplementation. | After 16 months of intervention
Patient survival with regards to high-dose vitamin D supplementation. | After 12 months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Hal Gunn, MD, Principal Investigator — University of British Columbia
Locations (1):
- InspireHealth, Vancouver, British Columbia, Canada

REFERENCES:
- See also: Related Info — http://www.inspirehealth.ca